CLINICAL TRIAL: NCT01946295
Title: Histamine H2 Antagonism as Adjuvant Therapy in Treatment Resistant Schizophrenia
Brief Title: Famotidine in Schizophrenia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jesper Ekelund (Other)
Collaborators: Karolinska Institutet (Other); Region Stockholm (Other Government); City of Helsinki (Other); Stanley Medical Research Institute (Other); Ahokas foundation, Finland (Unknown)
Responsible Party: Sponsor-Investigator, Jesper Ekelund, Professor, University of Helsinki
Organization: University of Helsinki (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-005513-40
Record Dates: First submitted 2013-08-23; First posted 2013-09-19 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Famotidine (Experimental): Famotidine 100mg x 2 orally
  Interventions: Drug: Famotidine
- Placebo (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Famotidine — 100mg x 2 p.o.
  Other Names: Famotidine Hexal; SUB07503MIG
  Arms: Famotidine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Objective of the trial is to study if famotidine add-on treatment is more effective than placebo add-on in reducing symptoms of schizophrenia among patients receiving insufficient response to ongoing antipsychotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* ICD-10 diagnosis of schizophrenia (F20.00-20.39, F20.5, F20.9) who have had the disorder for at least 5 years and who are on disability pension. (This means that their treatment response is not satisfactory and for the purpose of this study, the subjects are potentially treatment resistant).
* Clinical Global Impression (CGI) severity score of at least 3.
* No changes in schizophrenia treatment within 12 weeks before study inclusion.
* Written informed consent
* The subjects must fulfil schizophrenia criteria both according to DSM- IV (295.10, .20, .30, .60, .90) (American Psychiatric association) and the Research Diagnostic Criteria for schizophrenia (RDC) [40]. They must also have at least mild residual symptoms (CGI 3 points). The DSM-IV diagnosis will be verified by use of the SCID-I [41]. The DSM-IV is clearly the most commonly used in psychiatric research, so this is important to be able to generalize the findings. However, several previous studies have used the RDC, so to be able to compare the results, we will diagnose the patients according to both systems.
* Women of child-bearing age will be included only of they use adequate contraception, or if we can otherwise verify that the subject is not pregnant (s-HCG), the possibility of pregnancy is negligible (e.g. the personnel of the housing facility reports that the person has not had sexual relationships for years) and the subject approves to remain sexually abstinent for the duration of the study.

Exclusion Criteria:

* Epilepsy or a history of unclear seizures, stroke, Parkinson's disease, AIDS
* History of substance addiction or abuse within 3 months prior to enrolment.
* Individuals who are deemed at risk for aggressive behaviour or suicide
* If their laboratory tests, EKG or other clinical observation warrants exclusion, they will be excluded
* Women who are pregnant or breast-feeding subjects will not be included in the study.
* Patients with any serious unstable physical illness will also be excluded
* Patients who have been deemed to be legally incapacitated according to Finnish or Swedish law.
* Regular Uuse of H2-antagonists as prescribed by a physician.
* Known allergy to famotidine or any other component of interventional drug will be excluded.
* Ongoing treatment with clozapine and dixyrazine.
* Clinical condition "very much improved" or "much improved", assessed by CGI, during the placebo lead-in
* Renal insufficiency (P-creatinine not within normal range. Glomerular filtration rate <30 ml/min according to the Cockcroft-Gault formula. )
* Liver insufficiency (S-ALAT elevated more than 2-fold above the laboratory specific normal range)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Positive and Negative Syndrome Scale (PANSS) at 8 weeks | Rating at start of treatment (0 weeks) and at end of treatment (8 weeks)
  In addition PANSS ratings are done at screening, every two weeks during treatment and two weeks after end of treatment.

SECONDARY OUTCOMES:
Change from Baseline in Clinical Global Impression (CGI) scale at 8 weeks | Rating at start of treatment (0 weeks) and at end of treatment (8 weeks)
  In addition CGI ratings are done at screening, every two weeks during treatment and two weeks after end of treatment.
Change from Baseline in Calgary Depression Scale (CDS) at 8 weeks | Rating at start of treatment (0 weeks) and at end of treatment (8 weeks)
Change from Baseline in The Overall Anxiety Severity and Impairment Scale (OASIS)at 8 weeks | Rating at start of treatment (0 weeks) and at end of treatment (8 weeks)
Change from Baseline in CogState scores at 8 weeks | Rating at start of treatment (0 weeks) and at end of treatment (8 weeks)
  A standardized, language independent computerized battery of cognitive tests (CogState®). This battery has been validated and shown to be a sensitive indicator of mild impairments in the following cognitive domains: psychomotor speed, attention, working memory and episodic learning and memory.
Change from baseline in nightly sleep duration measured with actigraphy at 8 weeks | Measurement at start of treatment (0 weeks) and at end of treatment (8 weeks)
  Average nightly sleep duration of seven nights before and after intervention measured with an actigraph

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Ekelund, MD, PhD, Principal Investigator — University of Helsinki
Locations (6):
- Finland (4):
  - Helsinki University Central Hospital Psychiatry Centre, Helsinki
  - Helsinki University, Helsinki
  - Social services and Healthcare, City of Helsinki, Helsinki
  - Kellokoski Hospital, Hyvinkää
- Sweden (2):
  - Karolinska Institutet, Stockholm
  - Norra Stockholms Psykiatri, Stockholm County Council, Stockholm

REFERENCES:
- [Background] Meskanen K, Ekelund H, Laitinen J, Neuvonen PJ, Haukka J, Panula P, Ekelund J. A randomized clinical trial of histamine 2 receptor antagonism in treatment-resistant schizophrenia. J Clin Psychopharmacol. 2013 Aug;33(4):472-8. doi: 10.1097/JCP.0b013e3182970490. PMID 23764683